CLINICAL TRIAL: NCT04994522
Title: An Open-Label, Single-Dose Study to Investigate the Influence of Renal Impairment on the Pharmacokinetics of MK-6482
Brief Title: A Study of Belzutifan (MK-6482) in Participants With Renal Impairment (MK-6482-021)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-021; MK-6482-021 (Other: MSD)
Record Dates: First submitted 2021-08-02; First posted 2021-08-06 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease; Renal Impairment
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — belzutifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belzutifan in Participants with ESRD (Experimental): In period 1, participants with ESRD will receive a single, oral dose of belzutifan 120 mg on Day 1 after HD. In period 2, participants with ESRD will receive a single, oral dose of belzutifan 120 mg on Day 1 before HD. Each period is 4 days.
  Interventions: Drug: Belzutifan
- Belzutifan in Healthy Participants (Experimental): In period 1, healthy participants will receive a single, oral dose of belzutifan 120 mg on Day 1 of a 4-day period.
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — Three 40 mg tablets given as a single oral 120 mg dose.
  Other Names: MK-6482; PT2977; WELIREG

SUMMARY:
The primary purpose of this study is to compare the plasma pharmacokinetics (PK) of belzutifan (MK-6482) following a single oral 120 mg dose in participants with end stage renal disease (ESRD) before and after hemodialysis (HD) to each other and also to that of healthy matched control participants. This study will also evaluate the safety and tolerability of a single oral 120 mg dose of belzutifan in participants with ESRD and the extent of belzutifan removed by HD.

ELIGIBILITY:
Inclusion Criteria:

For Participants With Healthy Renal Function

* Is in good health based on the opinion of the investigator.
* Male participants agree to remain abstinent from heterosexual intercourse on a long-term basis or must agree to use contraception as instructed.
* Female participants must be of nonchildbearing potential.

For Participants With end stage renal disease (ESRD)

* With exception of the renal impairment, is in good health based on the opinion of the investigator.
* Has ESRD maintained on stable regimen of at least 3 times per week hemodialysis (HD) for at least 3 months prior to the initial administration of the study intervention.
* Male participants agree to remain abstinent from heterosexual intercourse on a long-term basis or must agree to use contraception as instructed.
* Female participants must be of nonchildbearing potential.

Exclusion Criteria:

For Participants With Healthy Renal Function

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Has a history of cancer (malignancy).
* Is positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV).
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Has received any non-live vaccine starting from 14 days prior to study intervention or is scheduled to receive any non-live vaccine through 30 days following study intervention (except coronavirus disease 2019 [COVID-19]).

Participants With ESRD

* Has a history of cancer (malignancy).
* Has required frequent emergent HD (≥3) within a year prior to the initial dose of study intervention.
* Is positive for HBsAg, hepatitis C antibodies, or HIV.
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Has received any non-live vaccine starting from 14 days prior to study intervention or is scheduled to receive any non-live vaccine through 30 days following study intervention (except COVID-19)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Orlando Clinical Research Center ( Site 0001), Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with end stage renal diseases (ESRD) and healthy matched control participants were recruited at a single study site in the United States.
Groups:
- Belzutifan in Participants With ESRD: In period 1, participants with ESRD received a single, oral dose of belzutifan 120 mg on Day 1 after hemodialysis (HD). In period 2, participants with ESRD received a single, oral dose of belzutifan 120 mg on Day 1 before HD. Each period is 4 days.
- Belzutifan in Healthy Participants: In period 1, healthy participants received a single, oral dose of belzutifan 120 mg on Day 1 of a 4-day period.
Period: Period 1
Arm/Group | Belzutifan in Participants With ESRD | Belzutifan in Healthy Participants
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Belzutifan in Participants With ESRD | Belzutifan in Healthy Participants
Started | 7 (Number started refers only to participants completing Period 1 volunteering to continue to Period 2.) | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Belzutifan in Participants With ESRD: In period 1, participants with ESRD received a single, oral dose of belzutifan 120 mg on Day 1 after HD. In period 2, participants with ESRD received a single, oral dose of belzutifan 120 mg on Day 1 before HD. Each period is 4 days.
- Total: Total of all reporting groups
Arm/Group | Belzutifan in Participants With ESRD | Belzutifan in Healthy Participants | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (8.48) | 55.5 (7.42) | 56.5 (7.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 0 | 4 | 4
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve of Belzutifan From Hour 0 to Infinity (AUC0-inf)
Description: AUC0-inf was defined as the area under the concentration-time curve of belzutifan from time zero to infinity. Blood samples collected predose and at multiple timepoints postdose were used to determine AUC0-inf of belzutifan in plasma.
Time Frame: Predose, and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, and 72 hours postdose
Population: All participants who are compliant with the study procedure and have available data considered sufficient to exhibit the effect of treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Groups:
- Belzutifan in Participants With ESRD Before HD (Period 2); Belzutifan in ESRD After HD (Period 1): In period 1, participants with ESRD received a single, oral dose of belzutifan 120 mg on Day 1 after HD. In period 2, participants with ESRD received a single, oral dose of belzutifan 120 mg on Day 1 before HD. Each period is 4 days.
Arm/Group | Belzutifan in Participants With ESRD Before HD (Period 2) | Belzutifan in ESRD After HD (Period 1) | Belzutifan in Healthy Participants
Number analyzed (Participants) | 7 | 8 | 6
ng•hr/mL | 17100 (91.3) | 21100 (91.3) | 18500 (41.4)

2. Primary Outcome: Area Under the Plasma Concentration Time Curve of Belzutifan From Hour 0 to 24 (AUC0-24)
Description: AUC0-24 was defined as the area under the concentration-time curve of belzutifan from time zero to 24 hours postdose. Blood samples collected predose and at multiple timepoints postdose were used to determine AUC0-24 of belzutifan in plasma.
Time Frame: Predose, and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Groups:
- Belzutifan in Participants With ESRD After HD (Period 1): In period 1, participants with ESRD received a single, oral dose of belzutifan 120 mg on Day 1 after HD. In period 2, participants with ESRD received a single, oral dose of belzutifan 120 mg on Day 1 before HD. Each period is 4 days.
Arm/Group | Belzutifan in Participants With ESRD Before HD (Period 2) | Belzutifan in Participants With ESRD After HD (Period 1) | Belzutifan in Healthy Participants
Number analyzed (Participants) | 7 | 8 | 6
ng•hr/mL | 10700 (50.5) | 12300 (50.7) | 13200 (30.7)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Belzutifan
Description: Cmax is the maximum concentration of belzutifan observed in plasma. Blood samples collected predose and at multiple timepoints postdose were used to determine Cmax of belzutifan in plasma.
Time Frame: Predose, and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Belzutifan in Participants With ESRD Before HD (Period 2) | Belzutifan in Participants With ESRD After HD (Period 1) | Belzutifan in Healthy Participants
Number analyzed (Participants) | 7 | 8 | 6
ng/mL | 1110 (44.0) | 907 (46.7) | 1300 (26.1)

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Belzutifan
Description: Tmax is the amount of time that belzutifan is present at the maximum concentration observed in plasma. Blood samples collected predose and at multiple timepoints postdose were used to determine Tmax of belzutifan in plasma.
Time Frame: Predose, and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Belzutifan in Participants With ESRD Before HD (Period 2) | Belzutifan in Participants With ESRD After HD (Period 1) | Belzutifan in Healthy Participants
Number analyzed (Participants) | 7 | 8 | 6
hour | 2.00 [1.00 to 3.00] | 4.00 [1.50 to 9.00] | 1.00 [0.50 to 3.00]

5. Primary Outcome: Apparent Terminal Half-life (t½) of Plasma Belzutifan
Description: t1/2 is defined as the time required to divide plasma concentration of belzutifan by half. Blood samples collected predose and at multiple timepoints postdose were used to determine the apparent terminal t1/2 of belzutifan in plasma.
Time Frame: Predose, and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Belzutifan in Participants With ESRD Before HD (Period 2) | Belzutifan in Participants With ESRD After HD (Period 1) | Belzutifan in Healthy Participants
Number analyzed (Participants) | 7 | 8 | 6
hour | 15.1 (68.1) | 17.1 (57.6) | 13.9 (20.9)

6. Secondary Outcome: Dialysis Clearance of Belzutifan Based on Plasma (CLD, Plasma)
Description: CLD, plasma is defined as a measure of the extent of belzutifan removed by HD. Blood samples collected at pre-dialysis and at multiple timepoints post-dialysis were used to measure the extent of belzutifan in plasma removal by HD.
Time Frame: Pre-dialysis, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, and 4 hours post-dialysis on Day 1 of Period 2 (Study Day ~12)
Population: Per protocol, CLD was measured in participants with ESRD who were treated with belzutifan before HD (Period 2). Participants in period 2 who are compliant with the study procedure and have available data considered sufficient to exhibit the effect of treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Belzutifan in Participants With ESRD Before HD (Period 2)
Number analyzed (Participants) | 7
mL/min | 78.4 (53.5)

7. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The percentage of participants who experienced an AE are reported.
Time Frame: Up to 32 days
Population: All participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Belzutifan in Participants With ESRD Before HD (Period 2) | Belzutifan in Participants With ESRD After HD (Period 1) | Belzutifan in Healthy Participants
Number analyzed (Participants) | 7 | 8 | 6
Percentage of Participants | 14.3 | 0.0 | 16.7

8. Secondary Outcome: Percentage of Participants Who Discontinue Study Intervention Due to an AE
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The percentage of participants who discontinue study intervention due to an AE are reported.
Time Frame: Up to 12 days
Population: All participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Belzutifan in Participants With ESRD Before HD (Period 2) | Belzutifan in Participants With ESRD After HD (Period 1) | Belzutifan in Healthy Participants
Number analyzed (Participants) | 7 | 8 | 6
Percentage of Participants | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to 32 days.
Description: All-Cause Mortality is reported for all allocated participants. Serious Adverse Events and Other Adverse Events are reported for all participants who received treatment. All adverse events that occurred after dosing are summarized. Every participant is counted a single time for each applicable adverse event.
Groups:
- Belzutifan in Participants With ESRD After HD (Period 2): In period 1, participants with ESRD received a single, oral dose of belzutifan 120 mg on Day 1 after HD. In period 2, participants with ESRD received a single, oral dose of belzutifan 120 mg on Day 1 before HD. Each period is 4 days.
Arm/Group | Belzutifan in Participants With ESRD Before HD (Period 2) | Belzutifan in Participants With ESRD After HD (Period 2) | Belzutifan in Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belzutifan in Participants With ESRD Before HD (Period 2) (N=7) | Belzutifan in Participants With ESRD After HD (Period 2) (N=8) | Belzutifan in Healthy Participants (N=6)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belzutifan in Participants With ESRD Before HD (Period 2) (N=7) | Belzutifan in Participants With ESRD After HD (Period 2) (N=8) | Belzutifan in Healthy Participants (N=6)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors (ICMJE) authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT04994522/Prot_SAP_000.pdf